CLINICAL TRIAL: NCT01211717
Title: The Effects of Orally Ingesting Branched Chained Amino Acids on Delayed Onset Muscle Soreness in Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Jerrold Petrofsky, PhD, Loma Linda University, School of Allied Health Professions
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5100233
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Type 2 Diabetes; Healthy Individuals
Keywords: Branched Chained Amino Acids; Delayed Onset Muscle Soreness; Diabetes; Muscle Damage
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Isoleucine; Leucine; Valine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Branched Chained Amino Acids (Experimental)
  Interventions: Dietary Supplement: Branched Chained Amino Acids
- Cellulose mix (Placebo Comparator)
  Interventions: Other: Cellulose Placebo mix

INTERVENTIONS:
Dietary Supplement: Branched Chained Amino Acids — Two doses of the Branched Chained Amino Acid supplement will be taken. The first dose will be taken 35 minutes before the intended exercise, and the other dose will be taken right after completing the exercise. The amount of the Branched Chained Amino Acid supplement administered to the subjects in the experimental group will vary from one person to the other but a total dose of 1 gram of BCAA per kilogram of lean body mass will be used. This dose will be divided in half and administered at the two specified occasions. The ratio of isoleucine, leucine, and valine will be 1:2.5:1 respectively
  Other Names: Isoleucine, Leucine, and Valine
  Arms: Branched Chained Amino Acids
Other: Cellulose Placebo mix — The control group will also take 2 doses, 1 before the exercise, and the other after completing the exercise. This dose will be divided in half and administered at the two specified occasions.
  Arms: Cellulose mix

SUMMARY:
The purpose of this study is to determine the effectiveness of the 3 Branched Chained Amino Acids (isoleucine, leucine, and valine) on treating Delayed Onset Muscle Soreness, a type of muscle pain which usually develops after exercising.

DETAILED DESCRIPTION:
Delayed Onset Muscle Soreness is a common painful sensation experienced by individuals who have been recently inactive and begin with an unaccustomed exercise protocol. Branched Chained Amino Acids have been found as a useful supplement for promoting muscle recovery following exercise; however the effects of this supplement have not been investigated amongst individuals with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* The subjects with diabetes must have been diagnosed with diabetes at least one year before the onset of the study
* At least 6 weeks of physical inactivity in the upper body
* BMI less than 40

Exclusion Criteria:

* For the Diabetics, hemoglobin A1c levels over 13
* Pregnant
* Have Cardiovascular diseases
* Have Hepatic diseases
* Are diagnosed with Rhabdomyolysis
* Recent upper limb injuries
* Upper limb neuropathy
* Blood Pressure levels over 140/90, or lower than 90/60
* Are on High doses of alpha or beta agonist/antagonists, and take any types of NSAID's, Cox 2 inhibitors, Calcium channel blockers, Pre-Gabalin's, or Pain reducers

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Measuring Pain, using the short form McGill pain questionnaire | 5 days following the initial exercise

SECONDARY OUTCOMES:
Measuring Muscle strength of the studied muscle | 5 days following the initial exercise

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Petrofsky, Doctoral PhD, Principal Investigator — Loma Linda University, School of Allied Health Professions
Locations (1):
- Loma Linda University, School of Allied Health Professions, Loma Linda, California, United States